CLINICAL TRIAL: NCT04021134
Title: The Effects of Allogeneic Simple Limbal Epithelial Transplantation
Brief Title: The Effects of Allogeneic SLET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904118RINB
Record Dates: First submitted 2019-07-03; First posted 2019-07-16 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-06

CONDITIONS: Limbal Stem-cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the effect of allogeneic SLET and re-epithelialization after allogeneic SLET.

DETAILED DESCRIPTION:
Simple limbal epithelial transplantation (SLET) was introduced in 2012 by Sangwan and coworkers to overcome the issues mainly related to the cost of a GMP-certified product and ease of surgical manipulations that al- lows use of smaller pieces of limbus from the contralateral eye (thus avoiding iatrogenic problems). A completely epithelialized, avascular and stable corneal surface was achieved by 6 weeks and was maintained in all recipient eyes at a mean follow-up of 9.2 ± 1.9 months. Best corrected visual acuity improved from worse than 20/200 in all recipient eyes before surgery to 20/40 or better in four (66.6%) eyes. None of the donor eyes developed any complications.Basu et al. reported autologous SLET on a population of 125 patients which included 65 adults and 60 children suffering from unilateral LSCD. 76% (95/125) of eyes maintained a successful outcome at final follow-up without progressive conjunctivalization, development of persistent epithelial defect, infection, or need for repeat SLET. Survival probability of 80% in adults and 72% in children after 1 year. So far, most of the reports have been about autoSLET, that is, the limbal explants are obtained from the unaffected eye of the same recipient, avoiding immune reaction at the later stage. Also, they demonstrated SLET had promising result both in adults and children. A study by Iyer and coworkers used alloSLET in early stages after ocular chemical injury to achieve rapid epithelialization. Instead of taking the biopsy from the recipient's healthy eye, they took it from a cadaveric donor and performed the SLET. Epithelialization and improved best corrected visual acuity and corneal phenotype were achieved at early stages; however, 7 of 18 eyes had a gradual failure of the allograft, and 5 eyes underwent subsequent limbal autograft. Symblepheron formation involving one to two quadrants was recorded in 3 eyes (16.7%). Visual rehabilitative procedures in the chronic phase of chemical injury, in most instances after alloSLET in the acute stage, did not require any keratoplasties. Unfortunately, most diseases causing limbal deficiency, e.g., surface burns (alkali/ thermal), Stevens-Johnson syndrome, contact lens-related epitheliopathy, and ocular cicatricial pemphigoid, tend to affect both eyes of a patient. Autologous SLET may not be applicable in patients with bilateral eyes involvement. In this study, the effect of allogeneic SLET will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 to 90 years old
2. The lesion eye has at least grade 2 limbal stem cell deficiency
3. The lesion eye has limbal stem cell deficiency causing recurrent corneal erosion and neovascularization ingrowth
4. The symptoms last for at least 6 months and do not improve with medication

Exclusion Criteria:

1. The symptoms improve spontaneously or with medication
2. Someone who can not be examined regularly after the operation
3. Poor prognosis
4. Severe lagophthalmos or trichiasis that has not been corrected
5. Ocular infection

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with limbal stem cell deficiency
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of patients with clinical success | 6 months
  Clinical success is defined as a completely epithelized, avascular, stable corneal surface. Failure was defined as a recurrence of fibrovascular pannus encroaching on the central cornea, frequent epithelial breakdown or persistent epithelial defects. Focal recurrences of pannus not progressing to the central cornea were not considered as failures and were evaluated separately.

SECONDARY OUTCOMES:
Best corrected visual acuity change | 6 months
  Best corrected visual acuity (BCVA) was measured with Snellen chart preoperatively and at 6 months after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, phD, Study Chair — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan, Republic of China
  - Department of Ophthalmology, National Taiwan University Hospital,, Taipei

IPD SHARING:
Plan to Share IPD: No
No IPD sharing in this study

REFERENCES:
- [Background] Borroni D, Wowra B, Romano V, Boyadzhieva M, Ponzin D, Ferrari S, Ahmad S, Parekh M. Simple limbal epithelial transplantation: a review on current approach and future directions. Surv Ophthalmol. 2018 Nov-Dec;63(6):869-874. doi: 10.1016/j.survophthal.2018.05.003. Epub 2018 May 22. PMID 29800578
- [Background] Iyer G, Srinivasan B, Agarwal S, Tarigopula A. Outcome of allo simple limbal epithelial transplantation (alloSLET) in the early stage of ocular chemical injury. Br J Ophthalmol. 2017 Jun;101(6):828-833. doi: 10.1136/bjophthalmol-2016-309045. Epub 2016 Oct 8. PMID 28407620